CLINICAL TRIAL: NCT02842632
Title: Evaluation of Simulator Training on Transesophageal Echocardiography (TEE) Performance in Anaesthesia Residents
Brief Title: Evaluation of Simulator Training on TEE Performance in Residents
Acronym: TEESimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulrike Weber (Other)
Responsible Party: Sponsor-Investigator, Ulrike Weber, Dr. Ulrike Weber, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1057/2016
Record Dates: First submitted 2016-07-15; First posted 2016-07-25 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A virtual teaching (Other): Group A will be introduced to the virtual TEE online (http://pie.med.utoronto.ca/TEE/)
  Interventions: Other: theoretical test; Other: practical test
- B simulator (Other): Group B will be introduced to the simulator (CAE Vimedix Simulator)
  Interventions: Other: theoretical test; Other: practical test
- C hands on OR (Other): group C will be introduced to the TEE training in the operation room.
  Interventions: Other: theoretical test; Other: practical test

INTERVENTIONS:
Other: theoretical test — The theoretical test is a multiple choice test which consists of 50 questions with 1 point per question (max. 50 points). It will be done before the teaching, after the 2 teaching sessions and 3 Months after the study
Other: practical test — The practical test is an evaluation of 11 basic perioperative TEE examination on the simulator (CAE Vimedix Simulator). Each view is evaluated on a scale of 0 to 10 according to predetermined criteria including image angle, overall clarity and visualization of 3 major anatomic structures pertinent to each view. Each view can receive a maximum score of 10 and each study a maximum of 109 (ME asc. aortic LAX has only 2 main structures). It will be done after the first and second teaching session, and 3 Months after the study.

SUMMARY:
Training in TEE is based on hands-on training in the operation room which is time consuming and therefore its use and experience is limited among anesthesiologists.

Recent studies demonstrate that simulation-based education is also superior to a conventional didactic system and superior to hands-on teaching in the OR in terms of theoretical knowledge in echocardiography. So far there is no study evaluating the study effect in obtaining the 11 basic TEE views as recommended by the American Society of Echocardiography (ASE) and the Society of Cardiovascular Anesthesiologists (SCA) between simulator training and training in the operation room in residents with no prior knowledge of echocardiography. The basic TEE examination focus on the 11 most relevant views.

Therefore the investigators want to assess if there is a difference in the study effect in obtaining the 11 basic TEE views and also in theoretical knowledge in 3 groups of residents with no prior knowledge of echocardiography:

the simulation group (CAE Vimedix Simulator), the hands-on OR group and the online group (http://pie.med.utoronto.ca/TEE/).

prospective randomized single-center study. The investigators want to include 51 anaesthesia residents (17 per group) in their first or second year of training with no prior knowledge of echocardiography in this randomized, Controlled single-centre study.

The investigators want to assess the pre- and post training scores of the theoretical multiple choice test and the practical test in all 3 groups. The multiple choice test consists of 50 questions with 1 point per question (max. 50 points) and the practical test is an evaluation of 11 basic perioperative TEE examination on the simulator (CAE Vimedix Simulator). Each view is evaluated on a scale of 0 to 10 according to predetermined criteria including image angle, overall clarity and visualization of 3 major anatomic structures pertinent to each view. Each view can receive a maximum score of 10 and each study a maximum of 109 (ME asc. aortic LAX has only 2 main structures). Further the time to adjust each view and the time to complete the basic TEE Examination will be assessed.

DETAILED DESCRIPTION:
The clinical utility of transesophageal echocardiography is increasingly recognized in perioperative medicine. However, training in TEE is based on hands-on training in the operation room which is time consuming and therefore its use and experience is limited among anesthesiologists.

Recent studies demonstrate that simulation-based education is also superior to a conventional didactic system and superior to hands-on teaching in the OR in terms of theoretical knowledge in echocardiography. So far there is no study evaluating the study effect in obtaining the 11 basic TEE views as recommended by the American Society of Echocardiography (ASE) and the Society of Cardiovascular Anesthesiologists (SCA) between simulator training and training in the operation room in residents with no prior knowledge of echocardiography. According tot he ASE and SCA the principal goal of the basic TEE examination is intraoperative monitoring. The basic TEE examination focus on the 11 most relevant views, which can enable anesthesiologists to diagnose general hemodynamic instability and its etiology in surgical patients and can in further consequence influence surgical outcome. The 11 basic TEE views are easier to remember and faster to obtain than a detailed 20 view standard examination.

Therefore the investigators want to assess if there is a difference in the study effect in obtaining the 11 basic TEE views and also in theoretical knowledge in 3 groups of residents with no prior knowledge of echocardiography:

the simulation group (CAE Vimedix Simulator), the hands-on OR group and the online group (http://pie.med.utoronto.ca/TEE/).

prospective randomized single-center study.

The investigators want to include 51 anaesthesia residents (17 per group) in their first or second year of training with no prior knowledge of echocardiography in this randomized, Controlled single-centre study.

Residents will be recruited by invitation for TEE training during their first or second year of residency in a large teaching hospital (AKH Wien).

The study will be conducted during 3 consecutive study days with a final exam (theoretical and practical on the third day).

The first study day will start with a lecture about the tested subjects, especially physical principles and heart anatomy. Then the students will complete a theoretical test (TT1) about basic knowledge for TEE, such as principles of ultrasonography, heart anatomy, indications as well as contraindications, patient safety and complications, probe manipulation and knowledge about basic pathologies (Severe hypovolemia, LV failure, RV failure, Tamponade, acute massive left-sided valvular regurgitation, circulatory arrest during resuscitation and after successful resuscitation.

Afterwards the participants will be randomised. After that, all students will get introduced to a protocol, which explains the examination process.

Group A will be introduced to the virtual TEE online (http://pie.med.utoronto.ca/TEE/), group B to the simulator (CAE Vimedix Simulator) and group C to the TEE training in the operation room.

From now on each student in group B and C will receive 2 practical sessions á 40 minutes within the next 2 weeks. Group A will study two times with the virtual TEE. The first practical session can be done on the first study day, the following one within 2 weeks and the final study day with the theoretical and practical test (TT2 and PT3) should be within 1 week after the second training session. All teaching sessions will start with a practical test (PT1 and PT2). This test will contain the 11 basic TEE views.

After the 2 teaching sessions all students will attend a second theoretical test (TT2) and a final practical tests (PT3). For the practical test the students should adjust and name the 11 basic TEE views within 10 minutes.

There will ba a follow up after 3 months with both a theoretical and a practical test (TT3 and PT4).

The investigators want to assess the pre- and post training scores of the theoretical multiple choice test and the practical test in all 3 groups. The multiple choice test consists of 50 questions with 1 point per question (max. 50 points) and the practical test is an evaluation of 11 basic perioperative TEE examination on the simulator (CAE Vimedix Simulator). Each view is evaluated on a scale of 0 to 10 according to predetermined criteria including image angle, overall clarity and visualization of 3 major anatomic structures pertinent to each view. Each view can receive a maximum score of 10 and each study a maximum of 109 (ME asc. aortic LAX has only 2 main structures). Further the time to adjust each view and the time to complete the basic TEE Examination will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* anaesthesia residents in their first or second year of clinical training

Exclusion Criteria:

* prior knowledge of echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in Score from the theoretical test | change from baseline to 1 day after training
  Change from Baseline test score at 1 day after training

SECONDARY OUTCOMES:
Change in score from practical test | change from baseline to 1 day after training
  Change from Baseline test score at 1 day after training

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Weber, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical university of vienna, General hospital of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No